CLINICAL TRIAL: NCT01433588
Title: Calmer: A Novel Approach for Treating Infant Pain
Brief Title: The Calmer Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's & Women's Health Centre of British Columbia (Other)
Responsible Party: Principal Investigator, Liisa Holsti, Associate Professor, Children's & Women's Health Centre of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CALMERP
Record Dates: First submitted 2011-09-09; First posted 2011-09-14 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Acute Pain
Keywords: Managing infant pain; 27 - 36+6 weeks gestation; Preterm infants
MeSH Terms: conditions — Acute Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calmer (Active Comparator): This therapeutic platform, called the Calmer interacts with the infant to help reduce stress to help promote better outcomes. It is being tested to see if it mimics Kangaroo care, maternal skin to skin, to help promote better health outcomes. Infants would be placed on it prior, during and after bloodwork to see if it elicits a favorable response.
  Interventions: Device: The Calmer
- Standard Care (Placebo Comparator): Standard of care during bloodwork is receiving a soother and facilitated tucking.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: The Calmer — This platform, called the Calmer, interacts with the infant to help reduce stress to help promote better outcomes. Infants can be placed on it for care to mimic Kangaroo Care, maternal skin to skin.
  Arms: Calmer
Other: Standard of Care — Infant would receive the standard of care for bloodwork, provided a soother and facilitated tucking.
  Arms: Standard Care

SUMMARY:
The purpose of this study is to see if the Calmer is more effective at managing acute pain in preterm infants in the neonatal intensive care than the current standard of care in the unit.

Hypothesis: While receiving treatment with Calmer, infants will show lower behavioral pain scores and lower heart rates, and more stable autonomic regulation as measured by heart rate variability indices, than infants given a soother plus facilitated tucking (standard of care) during routine blood collection.

DETAILED DESCRIPTION:
60 infants will be randomized to either receive the standard of care or the Calmer during a routine blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Stable infants admitted to the Neonatal Intensive Care Unit at Children's and Women's Health Centre of British Columbia (C&W)
* Preterm infants born at 27 to 36+6 completed weeks gestational age (GA) will be included
* GA is determined on the basis of the first day of the last menstrual period, early gestation ultrasonogram (in most cases) or best estimate based on neonatal examination
* Mothers must speak enough English to provide consent

Exclusion Criteria:

* Infants who have congenital anomalies, active, ongoing infection, or have undergone surgery
* Infants who have received pharmacological analgesics or sedatives within 72 hours of the assessment
* History of maternal abuse of controlled drugs and substances; blood collection that occurs beyond the 35th completed week (35 weeks + 6 days) GA
* Small for GA defined as a birth weight at least 2 standard deviations below mean for GA
* Higher order multiples (e.g. triplets)
* Infants in a cot

Ages: 27 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2014-10; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in Behavioral Indicators of Infant Pain (BIIP) Score | During the assessment period in the study, estimated to occur around one hour.
  The Behavioral Indicators of Infant Pain (BIIP) is a reliable and valid scale for assessing acute procedural pain in preterm infants.

SECONDARY OUTCOMES:
Secondary Outcome Measures: Heart Rate | During and after the assessment period in the study, estimated to be 6 hours.
  Heart rate will be recorded during the assessment period, one hour, to denote changes. Additionally, the heart rate will be recorded after the assessment period, for approximately 5 hours.
Secondary Outcome Measures: Heart Rate Variability | During and after assessment period in the study, estimated to be 6 hours.
  Heart rate variability during the assessment period will be recorded, monitored and reviewed for changes, estimated to occur over the course of an hour. Additionally, the heart rate variability will be recorded after the assessment period, for approximately 5 hours.
Secondary Outcome Measures: NIRS | During the assessment period in the study, estimated to occur over less than an hour.
  Brain blood oxy- and de-oxyhemoglobin, TSI, total hemoglobin, using near infra-red spectroscopy. During the assessment period in the study, estimated to occur around one hour.

CONTACTS AND LOCATIONS:
Overall Officials: Liisa Holsti, PhD, Principal Investigator — Developmental Neurosciences and Child Health, Child and Family Research Institute and Dept. of Occupational Science and Occupational Therapy, UBC
Locations (1):
- BC Children's and Women's Health Centre, Vancouver, British Columbia, Canada